CLINICAL TRIAL: NCT03468829
Title: A Randomized, Double-blind, Multicenter Study to Evaluate the Efficacy and Safety of ALX 0171 Versus Placebo, in Addition to Standard of Care, in Adults Who Have Undergone Hematopoietic Stem Cell Transplantation and Present With a Respiratory Syncytial Virus Respiratory Tract Infection
Brief Title: Efficacy and Safety of ALX-0171 in Adult Hematopoietic Stem Cell Transplant (HSCT) Recipients Who Present With Respiratory Syncytial Virus (RSV) Infection
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: ALX-0171 development program was stopped
Sponsor: Ablynx, a Sanofi company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALX0171-C204; 2017-003356-23 (EudraCT Number)
Record Dates: First submitted 2018-03-07; First posted 2018-03-19 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Respiratory Syncytial Virus Lower Respiratory Tract Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ALX-0171 Dose 1 (Experimental)
  Interventions: Biological: ALX-0171 Dose 1
- ALX-0171 Dose 2 (Experimental)
  Interventions: Biological: ALX-0171 Dose 2
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: ALX-0171 Dose 1 — Oral inhalation of ALX-0171 Dose 1 once daily for a maximum of 14 days
  Arms: ALX-0171 Dose 1
Biological: ALX-0171 Dose 2 — Oral inhalation of ALX-0171 Dose 2 once daily for a maximum of 14 days
  Arms: ALX-0171 Dose 2
Biological: Placebo — Oral inhalation of Placebo once daily for a maximum of 14 days
  Arms: Placebo

SUMMARY:
The primary objective of the study is to evaluate the antiviral effect and safety of inhaled ALX-0171 in adults diagnosed with respiratory syncytial virus (RSV) respiratory tract infection after hematopoietic stem cell transplantation (HSCT).

The secondary objective is to assess the clinical activity, pharmacokinetics (PK), virology, and immunogenicity of inhaled ALX 0171 in adults diagnosed with RSV respiratory tract infection after HSCT.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has received an HSCT using any conditioning regimen and for any underlying etiology (i.e., subject has received an autologous or allogeneic HSCT)
2. Subject is clinically diagnosed with RSV infection with new onset or acute worsening
3. Symptoms likely related to RSV infection have appeared within 5 days of screening and their severity requires initial or maintained hospitalization.
4. Documented RSV infection in the upper respiratory tract (URT)
5. Subject has:

   * Diagnosis of RSV lower respiratory tract (LRT) disease or
   * Diagnosis of RSV URT disease with high risk of progression to lower respiratory tract infection (LRTI)

Others as defined in the protocol

Exclusion Criteria:

1. Subject has clinically significant bacteremia or fungemia within 7 days of screening
2. Subject has clinically significant bacterial, fungal or viral pneumonia
3. Subject presents evidence of shock requiring intensive care unit (ICU) monitoring and/or vasopressor treatment
4. Subject requires or is expected to require invasive mechanical ventilation or intensive non-invasive respiratory support. Standard oxygen supplementation up to 6 L/minute is permitted provided it can be interrupted for the duration of study drug administration.

Others as defined in the protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-02 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Time-weighted average change from baseline in log10 RSV nasal viral load | From Day 1 to Day 7

SECONDARY OUTCOMES:
Safety as measured by the incidence of treatment-emergent (serious) adverse events | From Screening to Day 42
Nasal RSV load parameter: time to undetectable shedding | From Day 1 to Day 42
Clinical stabilization (defined as respiratory rate <25/minute and stable oxygen saturation >92% on room air for at least 12 hours) | From Day 1 to Day 42
Number of days without oxygen or with oxygen supplementation | From Day 1 to Day 42
Progression to lower respiratory tract (LRT) disease in subjects presenting with upper respiratory tract infection (URTI) at baseline | From Day 1 to Day 42
Concentration of ALX-0171 in serum | Day 1 to Day 14
  Measurement of ALX-0171 serum concentration at different time points from baseline until Day 14.
Immunogenicity as measured by the concentration of anti-ALX 0171 antibodies in serum | From Day 1 to Day 42

CONTACTS AND LOCATIONS:
Overall Officials: Ablynx Clinical Department, Study Director — Ablynx, a Sanofi company
Locations (5):
- Australia (2):
  - Investigator site, Darlinghurst
  - Investigator site, Westmead
- Investigator site, Leuven, Belgium
- Spain (2):
  - Investigator site 1, Valencia
  - Investigator site 2, Valencia

IPD SHARING:
Plan to Share IPD: No